Official Title: Enriched Environments: a Multi-level Integrative Medicine Intervention for Endometriosis

NCT#: NCT04179149

Date of last revision: 07/08/2019 INFORMED CONSENT

For women with endometriosis participating in the study on environmental enrichment and quality of life.

# Introduction and Purpose of the Study

Endometriosis is a condition that affects thousands of women and adolescents, usually during their reproductive years, causing severe pelvic pain that can become disabling and cause problems conceiving. Symptoms of endometriosis cause high levels of stress, frustration and poor quality of life in the affected women. The purpose of this study is to prove that enriching the environment with activities such as support groups, open spaces and learning stress management strategies can help patients with endometriosis to manage or reduce their pain and improve quality of life. To prove this, we propose to create an intervention called "environmental enrichment". This consists of participation in support groups that will meet once a month for six months in open places such as beaches, lakes, and parks. We hope that about 100 patients will participate in the study, which will be carried out in several phases.

In each session, participants will receive social support, and will also learn about new stress management strategies like yoga, relaxation, therapy with art, music and drama, and aromatherapy. The participants will answer questionnaires about their endometriosis related symptoms, and their physical and mental health. In addition, they will be asked to donate blood samples (to measure inflammatory molecules) and saliva (to measure stress markers). The participants will also have the opportunity to receive support during this period of time through social media platforms, such as WhatsApp and Facebook. With the information obtained during this study, we hope to demonstrate that complementary medicine strategies such as environmental enrichment can help improve the quality of life of women with endometriosis.

## **Explanation of the Procedures**

We will invite women with endometriosis to participate in the study through the social media page of the Puerto Rican Foundation for Endometriosis Patients (ENDOPR). Those interested in participating in the study will call the research team. During this call, several questions will be asked in order to asses if they meet the criteria to participate in the study. After orienting them and obtaining verbal consent to participate, patients will be assigned to one of two groups: the first group will receive the intervention in the first phase of the study, and the second group in the second phase. On the day of the first intervention, before beginning their participation in the study, participants must read and sign this document called Informed Consent.

Participation in this study is voluntary and involves the following:

- Partake in six (6) environmental enrichment sessions (one per month), which will be held at various points on the island such as La Guancha (Ponce), Baños de Coamo, Ponce Museum of Art, Lake Cerrillos (Ponce), among other open places.
- Complete a questionnaire about personal data, characteristics of the menstrual cycle, and symptoms, diagnosis and treatments of endometriosis (The EPhect questionnaire). This survey will be completed once and takes approximately 30 minutes to answer. The questionnaire will be sent by email for the participants to answer at their convenience.
- Answer several questionnaires to determine their levels of stress, depression, anxiety, quality of life, and observe how it relates to their experience as a patient with endometriosis:
  - 1. BAI measures anxiety levels (5 min)
  - 2. BDI measures levels of depression (5 min)
  - 3. Perceived Stress scale questions about events considered stressful in the past year (5 min)
  - 4. PROMIS-SF12 measures level of physical and mental health (10 min) (is completed electronically)
  - 5. EHP5 measures the impact of endometriosis on quality of life by asking how much the symptoms of endometriosis interfere with work, studies and daily activities. (5 min) (is completed electronically)
- Allow us access to audiotape participant-group communications during support groups and

observe interactions on social media platforms such as WhatsApp and Facebook. We will analyze the frequency of the interactions and the general topics of the discussions, without taking note of the identity of the participants.

- Allow us to contact the gynecologist of each participant to obtain clinical data confirming that
  the patient was diagnosed surgically with endometriosis, if treatment was received and the
  severity of the condition.
- Donate blood samples which will be used to measure the levels of inflammatory molecules and determine if the intervention can affect them in any way.
- Donate saliva samples to measure levels of stress hormones such as cortisol. The participants of the
  first group will complete these questionnaires and will donate a blood sample
  (approximately 4 tablespoons), during the interventions of months 1, 3 and 6, and 3 months after the
  interventions, adding a total of four (4) times.

The participants of the second group will complete these questionnaires and will donate a blood sample two (2) times, during educational activities scheduled in months 1 and 6 of the interventions. This group will then be invited to begin environmental enrichment interventions.

#### **Potential Benefits**

Participation in this study may not have any immediate or future benefits for the participants. It is possible for participants to benefit from learning stress management strategies, and exposure to open spaces and nature. In addition, during the interventions, participants will receive support from other patients and students of Clinical Psychology at the doctoral level. The participants will also receive support through social media groups on platforms like Facebook and WhatsApp. We hope the interventions implemented positively impact the quality of life of each participant and if deemed beneficial, will pave the way for future implementation of interventions such as environmental enrichment in the medical care of patients with endometriosis.

Participants will receive a \$ 20.00 gift card at each session to compensate for their time and expenses of transportation to the activities that are part of this study. The cost of all the materials, the resources and the entrance to the places where the sessions will take place will be covered by the researchers.

### **Risks or Discomforts**

We consider that participation in environmental enrichment sessions does not entail mayor risks. There is a small risk that participants may feel uncomfortable with some of the questions asked, especially those that are included in the questionnaires that measure stress, anxiety and depression. To minimize this risk, the questionnaires will be completed in the presence of a trained professional (students of Clinical Psychology at the doctoral level, under the supervision of licensed Clinical Psychologists). If any concern for the general welfare and mental health of the participants arises, 1) immediate attention and / or 2) referral will be provided for services in psychological services clinics (for example, the PHSU Wellness Clinic). Additionally, all participants will be provided with phone numbers of local clinics that provide psychological and crisis management services (such as the PAS hotline).

The risks associated with donating blood samples are considered minimal, since they are not greater than the common blood samples taken in clinical laboratories. There is always a minimal risk of discomfort, infection or bruising caused by the needle, but this risk will be minimal since the samples will be taken by trained personnel. The donation of saliva samples does not involve any risk.

There is a risk that your personal and clinical information may be seen by an unauthorized person. We will make this risk very small by keeping all the information encoded with a number (never with your name) and stored in a secure place with restricted access.

## Confidentiality

All data obtained in this study will be treated with strict confidentiality, as required by the federal HIPAA law. A numerical code will be placed on all the questionnaires and data with the purpose of protecting the privacy of the participants. The document containing the assigned names and codes

will be kept locked in the office of Dr. Flores. Only Dr. Idhaliz Flores and doctoral students of the PhD Program of Clinical Psychology and researchers of the study will have access to the data that identify the participants. Only coded data without information identifying the participants will be shared with the study collaborators. All the information obtained from the participants, including the transcripts of the support group meetings, will be kept on a computer with restricted access, using a computer program protected by security codes (passwords). The results of this study that are presented at scientific conferences or that are published will not include information that can identify the participants.

## Withdrawal from the Study

Participation in this study is voluntary. Patients can freely decide not to participate or withdraw at any time without this representing any consequence to their health care. In the case of withdrawal from the study, no additional information or samples will be obtained. The information of the withdrawing participant will not be included in the final conclusions of the investigation.

#### Questions

For questions about this study, you can contact Dr. Idhaliz Flores, principal investigator of the Ponce Research Institute (PRI), at 787-840-2575 ext. 2206. For questions about rights as a participant in this research, you can contact Dr. Simón Carlo, director of the Institutional Review Board (IRB) of the PRI at PO Box 7004, Ponce, PR or 787-840-2575 ext. 2158

\_\_\_\_\_\_

If after reading this information you agree to participate in the study, please sign the informed consent that is presented below:

## **Informed Consent**

I understand all the information provided in this document and I have been informed about the risks and benefits of this investigation. I have been assured that the researchers in this study will be available to answer any questions I may have. I understand that I can freely choose not to participate in this research and that I may withdraw my participation at any time, even after signing this form, and that this will not have any consequence on my medical care. By signing this form, I am consenting to participate in this study, clearly understanding the information provided here. I will receive a copy of the signed form for my records.

| PARTICIPANT'S NAME: | DATE: _ |
|--------------------------------|---------|
| PARTICIPANT'S SIGNATURE: | |
| NAME OF THE INVESTIGATOR: | DATE: |
| SIGNATURE OF THE INVESTIGATOR: | |

### **CONSENTIMIENTO INFORMADO**

Para mujeres con endometriosis participantes en el estudio sobre enriquecimiento ambiental y calidad de vida

### Introducción y Propósito del Estudio

La endometriosis es una condición que afecta a miles de mujeres y adolescentes, generalmente durante sus años reproductivos, causándoles dolor pélvico severo que puede llegar a ser incapacitante y causar problemas para quedar embarazadas. Los síntomas de la endometriosis causan altos niveles de estrés, frustración y pobre calidad de vida en las mujeres afectadas. El propósito de este estudio es probar que enriquecer el ambiente con actividades como grupos de apoyo, espacios abiertos y aprender estrategias de manejo de estrés puede ayudar a las pacientes con endometriosis a manejar o disminuir el dolor y a mejorar su calidad de vida. Para probar esto, proponemos crear una intervención llamada "enriquecimiento ambiental". Esta consiste en la participación en grupos de apoyo que se reunirán una vez al mes durante seis meses en lugares abiertos como playas, lagos, y parques. Esperamos que cerca de 100 pacientes participen en el estudio, el cual se llevará cabo en varias fases.

En cada sesión, las participantes recibirán apoyo social, y además aprenderán sobre nuevas estrategias de manejo de estrés como yoga, relajación, terapia con arte, música y drama, y aromaterapia. Las participantes contestarán cuestionarios sobre sus síntomas relacionados con la endometriosis, su salud física y mental. Además, se les pedirá que donen muestras de sangre (para medir moléculas inflamatorias) y de saliva (para medir marcadores de estrés). Las participantes también tendrán la oportunidad de recibir apoyo durante este periodo a través de plataformas sociales como Whatsapp y Facebook. Con la información obtenida durante este estudio esperamos demostrar que estrategias de medicina complementaria como el enriquecimiento ambiental pueden ayudar a mejorar la calidad de vida de las mujeres con endometriosis.

### Explicación de los Procedimientos

Invitaremos a mujeres con endometriosis a participar a través de medios de comunicación social de la <u>Fundación Puertorriqueña de Pacientes con Endometriosis</u> (ENDOPR). Aquellas interesadas en participar en el estudio llamarán al equipo de investigación. Durante esta llamada, se harán varias preguntas para evaluar si cumplen con los requisitos para participar en el estudio. Luego de la orientación, se obtendrá consentimiento verbal para participar de aquellas que cumplen con los requisitos. Las pacientes serán asignadas a uno de dos grupos: el primer grupo recibirá la intervención en los primeros seis meses del estudio (primera fase), y el segundo grupo en la segunda fase que se llevará a cabo en los meses subsiguientes. El día de la primera intervención, antes de comenzar su participación en el estudio, las participantes deben leer y firmar este documento llamado **Consentimiento Informado**.

La participación en este estudio es **voluntaria** y conlleva lo siguiente:

- Participar en seis (6) sesiones de enriquecimiento ambiental (una por mes), que se llevarán a cabo en diversos puntos de la isla como La Guancha (Ponce), Baños de Coamo, Museo de Arte de Ponce, Lago Cerrillos (Ponce), entre otros lugares abiertos.
- Completar un cuestionario con datos personales, características del ciclo menstrual, y síntomas, diagnóstico y tratamientos de endometriosis. Este cuestionario se completará una sola vez y toma aproximadamente 30 minutos en contestarse. El cuestionario se enviará por correo electrónico para que las participantes lo contesten a su conveniencia.
- Contestar varios cuestionarios para determinar sus niveles de estrés, depresión, ansiedad, satisfacción sexual, impacto en la calidad de vida, y sobre su experiencia como paciente de endometriosis:
  - 1. BAI mide los niveles de ansiedad (5 min)
  - 2. BDI mide los niveles de depresión (5 min)
  - 3. Perceived Stress Scale pregunta sobre eventos considerados estrésicos en el pasado año (5 min)
  - 4. PROMIS/SF12 mide nivel de salud física y mental (10 min) (se completa electrónicamente)
  - 5. EHP5 mide el impacto de la endometriosis en la calidad de vida al preguntar cuánto los síntomas de la endometriosis interfieren con el trabajo, estudios y actividades diarias. (5 min) (se completa electrónicamente)
- Permitirnos acceso a grabar las discusiones durante los grupos de apoyo y a observar las comunicaciones del grupo de participantes en plataformas sociales como Whatsapp y Facebook. Analizaremos la frecuencia de las interacciones y los temas generales de las discusiones, sin tomar nota de la identidad de las participantes.
- Permitirnos comunicarnos con su ginecólogo para obtener datos clínicos que confirmen que la paciente fue diagnosticada guirúrgicamente con endometriosis, si se recibió tratamiento y la gravedad de la condición.
- Donar muestras de sangre las cuales se usarán para medir los niveles de moléculas inflamatorias y determinar si la intervención puede afectarlas de alguna manera.
- Donar muestras de saliva para medir los niveles de hormonas de estrés como el cortisol.

Las participantes del primer grupo completarán estos cuestionarios y donarán una muestra de sangre (aproximadamente 4 cucharadas), durante las intervenciones de los meses 1, 3 y 6, y a los 3 meses de finalizadas las intervenciones, sumando un total de **cuatro (4) veces** 

Las participantes del segundo grupo completarán estos cuestionarios y donarán una muestra de sangre <u>dos (2)</u> <u>veces</u>, durante actividades educativas programadas en los meses 1 y 6 de las intervenciones. Seguidamente este grupo comenzará las intervenciones de enriquecimiento ambiental según descrito arriba para el grupo experimental.

#### **Beneficios Potenciales**

La participación en este estudio podría no tener ningún beneficio inmediato ni futuro para las participantes. Es posible que para las participantes sea un beneficio aprender estrategias de manejo de estrés, y la exposición a espacios abiertos y a la naturaleza. Además, durante las intervenciones, las participantes recibirán apoyo de otras pacientes y estudiantes de Psicología Clínica a nivel doctoral. Los participantes también recibirán apoyo a través de grupos de medios sociales en plataformas como Facebook y WhatsApp. Esperamos que las intervenciones implementadas tengan un impacto positivo en la calidad de vida de cada participante y, si se consideran beneficiosas, allanarán el camino para la implementación futura de intervenciones como el enriquecimiento ambiental en la atención médica de pacientes con endometriosis.

Las participantes recibirán \$20.00 en cada sesión para compensar su tiempo y gastos de transportación a las actividades que son parte de este estudio. El costo de todos los materiales, los recursos y la entrada a los lugares donde se llevarán a cabo las sesiones estarán cubiertos por los investigadores.

### Riesgos o Incomodidades

Consideramos que la participación en las sesiones de enriquecimiento ambiental no conlleva riesgos mayores. Existe un pequeño riesgo de que las participantes puedan sentirse incómodas con algunas de las preguntas que se les hagan, especialmente aquellas que se incluyen en los cuestionarios que miden estrés, ansiedad y depresión. Para minimizar este riesgo, los cuestionarios se completarán en presencia de un profesional entrenado (estudiantes de Psicología Clínica a nivel doctoral, bajo la supervisión de Psicólogos Clínicos con licencia). Si surgiera cualquier preocupación por el bienestar general y de salud mental de las participantes, se proveerá 1) atención inmediata y/o 2) referido para servicios en clínicas de servicios psicológicos (por ejemplo el Wellness Clinic de PHSU). Adicionalmente, se les proveerá a todas las participantes los números de teléfono de clínicas locales que brindan servicios psicológicos y apoyo en crisis (ej. La Línea de crisis PAS).

Los riesgos asociados a donar muestras de sangre son considerados mínimos, ya que no son mayores a las muestras comunes de sangre tomada en los laboratorios clínicos. Siempre hay un riesgo mínimo de molestia, infección o formación de hematomas causados por la aguja, pero este riesgo será mínimo ya que las muestras serán tomadas por personal entrenado. La donación de muestras de saliva no conlleva riesgo alguno.

Existe el riesgo de que su información personal y clínica puedan ser vistas por personas no autorizadas. Haremos este riesgo muy pequeño al mantener toda la información codificada con un número (nunca con su nombre) y guardada en un lugar seguro con acceso restringido.

#### Confidencialidad

Todos los datos que se obtengan en este estudio se tratarán con estricta confidencialidad, tal y como lo requiere la ley federal HIPAA. Se colocará un código numérico a todos los cuestionarios y los datos con el propósito de proteger la privacidad de las participantes. Las transcripciones de los grupos de apoyo y las anotaciones de las intereacciones de los Chat Rooms serán obtenidas sin referencia a nombres de las participantes. El documento que contenga los nombres y códigos asignados se mantendrá bajo llave en la oficina de la Dra. Flores. Únicamente la Dra. Idhaliz Flores y estudiantes doctorales del Programa PhD de Psicología Clínica e investigadores del estudio tendrán acceso a los datos que identifican a las participantes. Solamente datos codificados sin información que identifique a las participantes serán compartidos con los colaboradores del estudio para propósito de análisis. Toda la información que se obtenga de las participantes, incluyendo las transcripciones de los grupos de apoyo, se mantendrán en una computadora con acceso restringido, utilizando un programa de computadora protegido por códigos de seguridad (passwords). Los resultados de este estudio que se presenten en conferencias científicas o que se publiquen no incluirán información que pueda identificar a las participantes.

# Retiro del Estudio

La participación en este estudio es **voluntaria**. Las pacientes pueden decidir libremente no participar o retirarse en cualquier momento sin que esto represente ninguna consecuencia al cuidado de su salud. En el caso de retiro del estudio, no se obtendrá información ni muestras adicionales. La información de la participante que se retira no se incluirá en las conclusiones finales de la investigación.

## Preguntas

| Para preguntas acerca de este estudio, puedes contactar a la Dra. Idhaliz Flor del Ponce Research Institute (PRI), al 787-840-2575 ext. 2206. Para preguntas esta investigación, puedes contactar al Dr. Simón Carlo, director de el Comité de inglés) del PRI al PO Box 7004, Ponce, PR o al número de teléfono 840-2575 ext. | sobre derechos como participante de<br>e Revisión Institucional (IRB, siglas en |
|---|---|
| Si después de haber leído esta información estás de acuerdo con participar en e miento informado que se presenta a continuación: | el estudio, firma por favor el consenti- |
| Consentimiento Informado: | |
| Entiendo toda la información provista en este documento y he sido informada sobre los riesgos y beneficios de esta investigación. Se me ha asegurado que los investigadores en este estudio estarán disponibles para contestar cualquier pregunta que yo pueda tener. Entiendo que puedo elegir libremente no participar en esta investigación y que puedo retirar mi participación en cualquier momento, aún después de firmar este formulario, y que esto no tendrá ninguna consecuencia en mi cuidado médico. Al firmar este formulario, estoy consintiendo a participar en este estudio, entendiendo claramente la información aquí provista. Recibiré una copia del formulario firmado para mis expedientes. | |
| NOMBRE DEL PARTICIPANTE: | FECHA: |
| FIRMA DEL PARTICIPANTE: | |

NOMBRE DEL INVESTIGADOR(A): \_\_\_\_\_ FECHA: \_\_\_\_

FIRMA DEL INVESTIGADOR(A): \_\_\_\_\_